CLINICAL TRIAL: NCT00186589
Title: 90Y-Ibritumomab Tiuxetan and Autologous Hematopoietic Cell Infusion Followed by High Dose Chemotherapy and Autologous Transplantation for Relapsed or Resistant Non-Hodgkin's Lymphoma
Brief Title: 90Y-IBRITUMOMAB Tiuxetan and AHCI With HD Chemotherapy and Autologous Transplantation for Relapsed or Resistant NHL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Biogen (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sandra Jeane Horning, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT134; 80109; BMT134; NCT00186589
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2010-10

CONDITIONS: Lymphoma, Non-Hodgkin; Blood and Marrow Transplant (BMT)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan

INTERVENTIONS:
Drug: 90Y Ibritumomab tiuxetan

SUMMARY:
To test a new way to approach hematopoietic stem cell transplantation for Relapsed or Resistant Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
This is a single center phase I dose escalation trial of a single course of IDEC-Y2B8 (90Y-ibritumomab tiuxetan, Zevalin) with autologous peripheral blood progenitor cell infusion followed by high dose chemotherapy and AHCT for patients with relapsed or refractory B-cell NHL. In step one, an imaging dose of IDEC-In2B8 (111In- ibritumomab tiuxetan, Zevalin) will be followed one week later by IDEC-Y2B; both will be preceded by an infusion of 250 mg/m2 rituximab. Imaging will be done immediately (within 1 hr), at 4 - 6 hours and at 1, 3, and 6 days after 90Y-ibritumomab tiuxetan.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria -- Step 1

4.1 Histologically proven, recurrent or refractory, CD20+ B-cell NHL reviewed at SUMC.

4.11 The definition of recurrent disease is: previous partial response (PR) or complete response (CR) to treatment followed by disease progression.

4.12 The definition of refractory disease is: failure to achieve a PR or CR with or progression during primary induction therapy or subsequent salvage therapy. Patients who respond to treatment but progress within 60 days will also be considered refractory.

4.13 CD20 expression may be determined by immunohistochemistry or flow cytometry. Whenever possible, confirmation of CD20+ status should be made on current, active disease.

4.14 The definition of NHL will be made by SUMC pathologists using the World Health Organization Classification of Hematopoietic and Lymphoid Tissues (Appendix A).

4.15 The diagnosis should be made by excisional biopsy whenever possible. Biopsy of refractory or recurrent disease is preferred but fine needle aspirate with supportive morphology and immunohistochemistry is acceptable. Paraffin tissue for tissue array studies will be sought for every patient.

4.2 Age 18-70 years

4.21 Age will be based on actual date of birth.

4.22 Pediatric patients are not eligible for this study because they are transplanted in a separate dedicated unit with their own protocols.

4.3 ECOG performance status 0-2 (Appendix B)

4.4 Computerized tomography scans of the chest, abdomen and pelvis within 4 weeks of registration. Assessment of response to last chemotherapy prior to registration is mandatory.

4.41 Response will be assessed according to the international consensus criteria (Cheson et al. J Clin Oncol 17:1244, 1999)

4.42 Standard definitions of the chest, abdomen and pelvis will be used for radiographic studies.

4.5 Gallium scan or PET scan determination of disease within 4 weeks of registration is highly recommended.

4.51 Gallium or PET scans will be whole body scans

4.6 Bone marrow biopsy and cytogenetic analysis within 8 weeks of registration. Patients must have no or <25% involvement of the intratrabecular bone marrow cellularity by NHL.

4.7 Adequate (> 4 x 10^6/kg CD34+) peripheral blood progenitor cells collected by apheresis.

4.8 Women of child-bearing potential and sexually active males are strongly advised to use an accepted and effective method of birth control.

4.9 No chemotherapy other than corticosteroids should be administered within 4 weeks of the initiation of protocol therapy.

4.10 Pretreatment absolute neutrophil count > 1000/mm^3 and platelet count > 150,000/ mm^3.

4.11 Patients must have a pretreatment serum bilirubin < 2 x the institutional ULN, transaminases < 2 x the institutional ULN, a serum creatinine < 2 x the institutional ULN and measured or estimated creatinine clearance > 60 cc/min by the following formula (all tests must be performed within 28 days prior to registration):

Estimated Creatinine Clearance = (140 age)X WT(kg) X 0.85 if female X creatinine (mg/dl)

4.12 Patients must have an EKG within 42 days prior to registration that shows no significant abnormalities that are suggestive of active cardiac disease.

4.13 Patients must have a radionuclide ejection fraction >45% within 42 days of registration.

4.14 Patients must have a corrected diffusion capacity 70% or greater.

4.15 Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Inclusion Criteria -- Step 2

4.30 Absolute neutrophil count recovery to > 1000/mm^3 and platelet recovery count to > 100,000/ mm^3.

4.31 Corrected diffusing capacity > 60%.

4.32 Resting ejection fraction of > 45%.

4.33 Serum bilirubin < 2, SGOT (AST) < 2 x ULN, SGPT (ALT) < 2 x ULN. Creatinine < 2 x the ULN and measured or estimated creatinine clearance > 60 cc/min. Exclusion Criteria:Exclusion Criteria - Step 1

4.16 Patients with known allergy to etoposide or a history of Grade 3 hemorrhagic cystitis with cyclophosphamide are not eligible.

4.17 No prior malignancy is allowed except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other cancer for which the patients has been disease-free for five years.

4.18 Patients known to be human immunodeficiency virus (HIV)-positive are ineligible because the concern for opportunistic infection and hematologic reserve are considered to be significantly greater in this population. The antibody test for HIV must be performed within 42 days of registration.

4.19 Patients requiring therapy for coronary artery disease, cardiomyopathy, dysrhythmia, or congestive heart failure are not eligible.

4.20 Pregnant or breast-feeding women are ineligible due to the known birth defects associated with the treatments used in this study.

4.21 Patients with prior radiotherapy to >25% of the active marrow are excluded.

4.22 Patients treated previously with radioimmunotherapy are excluded.

4.23 Patients with pleural effusion or ascites are excluded.

4.24 Patients may have received prior rituximab but not within the past 4 weeks.

4.25 Patients with prior autologous transplantation are ineligible.

4.26 Patients with CNS disease are ineligible.

Exclusion Criteria - Step 2

4.33 Drop in diffusing capacity of >25% from study entry.

4.34 Drop in resting ejection fraction > 20%.

4.35 Failure to recover peripheral blood counts (ANC > 1000/mm^3 and platelet recovery count to > 100,000/mm^3 within 4 weeks after radioimmunotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Complete Response | completed

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jeane Horning, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States